CLINICAL TRIAL: NCT03176641
Title: Efficacy of Platelet-rich Plasma on Meniscus Repair- a Randomized Controlled Trial
Brief Title: Platelet-rich Plasma for Meniscus Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Superintendent, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RA-16027-RD-105063
Record Dates: First submitted 2017-04-13; First posted 2017-06-05 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Platelet-Rich Plasma; Knee Injuries; Meniscus Disorder
Keywords: Platelet-Rich Plasma; Meniscus; Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRP group (Active Comparator): 30 patients will receive autologous platelet-rich plasma gel during meniscus repair surgery.
  Interventions: Other: platelet-rich plasma
- Control group (Placebo Comparator): 30 patients will receive meniscus repair surgery only.
  Interventions: Other: control

INTERVENTIONS:
Other: platelet-rich plasma — Autologous platelet-rich plasma gel applied during meniscus repair surgery
  Arms: PRP group
Other: control — Meniscus repair surgery only
  Arms: Control group

SUMMARY:
This study aims to evaluate the effect of platelet-rich plasma (PRP) on meniscus injury by comparing the imaging and clinical outcomes between patients receiving PRP with meniscus repair surgery and those receiving meniscus repair surgery only.

DETAILED DESCRIPTION:
Damage to meniscal tissue is challenging for orthopedic surgeons because of the absence of healing at the avascular zone. Additionally, the accelerated degeneration of articular cartilage and increased rate of knee osteoarthritis that can occur following a meniscal injury. Platelet-rich plasma (PRP) is a fraction of plasma that contains platelets and multiple growth factors concentrated at high level. Because activated platelets have the potential to release growth factors, PRP has been clinically used to accelerate wound healing and tissue regeneration in orthopedic and oral surgery. Several in vivo and in vitro studies have reported favorable outcomes of PRP on meniscal repair; however, the clinical results varied between studies.This clinical trial will investigate the effect of PRP on on meniscus injury. Eligible patients will be randomly assigned to receive PRP with meniscus repair surgery or to receive meniscus repair surgery only. The postoperative imaging and clinical outcomes will be compared and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 60 years
* With diagnosis of meniscus injury
* With indications of meniscus repair surgery

Exclusion Criteria:

* Multiple ligaments injury
* with prior history of knee surgery
* Cancer patients
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
3-month postoperative knee function evaluated by IKDC | 3-month postoperative
  Knee function is evaluated using International Knee Documentation Committee (IKDC) score.

SECONDARY OUTCOMES:
6-month postoperative knee function evaluated by IKDC | 6-month postoperative
  Knee function is evaluated using International Knee Documentation Committee (IKDC) score.
12-month postoperative knee function evaluated by IKDC | 12-month postoperative
  Knee function is evaluated using International Knee Documentation Committee (IKDC) score.
3-month postoperative knee pain evaluated by VAS | 3-month postoperative
  Pain level is evaluated using visual analogue scale (VAS).
6-month postoperative knee pain evaluated by VAS | 6-month postoperative
  Pain level is evaluated using visual analogue scale (VAS).
12-month postoperative knee pain evaluated by VAS | 12-month postoperative
  Pain level is evaluated using visual analogue scale (VAS).
Percentage of patients with healed meniscus 6-month postoperative | 6-month postoperative
  Healing of meniscus is evaluated by MRI
Percentage of patients with healed meniscus 12-month postoperative | 12-month postoperative
  Healing of meniscus is evaluated by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No